CLINICAL TRIAL: NCT04692376
Title: Mesenchymal Stem Cell for Treatment of Chronic Graft-versus-host Disease After Allogenetic Hematopoietic Stem Cell Transplantation
Brief Title: MSC for Treatment of cGVHD After Allo-HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-sen University (Other); Army Medical University, China (Other); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-cGVHD-2020
Record Dates: First submitted 2020-12-26; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Chronic Graft-versus-host Disease
Keywords: Hematopoietic Stem Cell Transplantation; Chronic Graft-versus-host disease; Mesenchymal Stem Cells
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Glucocorticoids; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSCs group (Experimental): MSCs group refers to treatment with mesenchymal stem cells (1×10^6 cells/kg, intravenously) weekly for 8 doses. Besides, glucocorticoids and cyclosporine (CsA) will be used for treatment concurrently.
  Interventions: Biological: Mesenchymal stem cells; Drug: Glucocorticoids; Drug: cyclosporine
- Control group (Active Comparator): Glucocorticoids and CsA will be used for treatment.
  Interventions: Drug: Glucocorticoids; Drug: cyclosporine

INTERVENTIONS:
Biological: Mesenchymal stem cells — Mesenchymal stem cells (MSCs) will be intravenously infused via a central venous catheter(at a dose of 1×10^6 cells/kg, over 15 mins) weekly. MSCs will be administrated for 8 doses.
  Arms: MSCs group
Drug: Glucocorticoids — Glucocorticoids (i.e. Methylprednisolone) will be used with an initial dose of 1mg/kg.
Drug: cyclosporine — Cyclosporine (CsA) will be used with an initial dose of 2.5mg/kg/d and adjusted according to the concentration of CsA. The targeted concentration is 200-300 ng/Ml.

SUMMARY:
The purpose of this study is to evaluate the efficacy of mesenchymal stem cells in patients with chronic graft-versus-host disease.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation(allo-HSCT) can cure many hematologic diseases. Although great progress has been made in the prevention and treatment of side effects associated with transplantation,chronic graft-versus-host disease(cGVHD) remains an important complication that occurs in about 50% patients. The mortality of cGVHD and its complication could reach up to 50%,and cGVHD seriously influence the quality of life. At present, the first line treatment of cGVHD remains in discussion.

Mesenchymal stem cells (MSCs) are a form of multipotent adult stem cells that can be isolated from bone marrow (BM), adipose tissue, and cord blood. Clinical applications of human MSCs are evolving rapidly with goals of improving hematopoietic engraftment, preventing and treating GVHD after allo-HSCT and so on. However, the efficacy of treatment of cGVHD remains undetermined.

In the present study, the investigators will prospectively evaluate the efficacy and safety of ex-vivo-expanded MSCs in treating patients with cGVHD.

ELIGIBILITY:
Inclusion Criteria:

* A patient age of 18-65 years
* Recipients of allogeneic hematopoietic stem cell transplantation Patients with moderate/ severe cGVHD without systemic treatment
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Primary disease relapse
* Expected lifetime less than 3 months
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2021-01-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 weeks after the first dose of MSCs
  Overall response rate （ORR）includes complete response (CR) and part response (PR).

SECONDARY OUTCOMES:
OS | 1 year after the first dose of MSCs
  Overall survival (OS)
DFS | 1 year after the first dose of MSCs
  Disease-free survival (DFS)
Response rate | 4 weeks after the first dose of MSCs
EBV DNA-emia | 1 year after the first dose of MSCs
  EBV DNA-emia refers to detection of EBV DNA in peripheral blood via PCR.
CMV DNA-emia | 1 year after the first dose of MSCs
  CMV DNA-emia refers to detection of CMV DNA in peripheral blood via PCR.
PGF | 1 year after the first dose of MSCs
  Poor graft function (PGF) refers to a slow or incomplete recovery of blood cell counts (ANC ≤0.5x10^9/L and PLT ≤20x10^9/L) by +28 days after allo-HSCT or a fall in blood cell counts to levels fulfilling the diagnostic criteria for PGF after successful and prompt hematopoietic engraftment.

CONTACTS AND LOCATIONS:
Overall Officials: Qi-fa Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China